CLINICAL TRIAL: NCT04498624
Title: Vitrectomy and Inverted Flap or Internal Limiting Membrane Peeling in Small Full Thickness Macular Holes
Brief Title: Inverted Flap Versus Internal Limiting Membrane Peeling in Small Full Thickness Macular Holes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Michele Reibaldi, Prof., University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0062156
Record Dates: First submitted 2020-07-22; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Full Thickness Macular Hole
Keywords: Full thickness macular hole; Vitrectomy; Inverted flap; Internal limiting membrane peeling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inverted flap (Active Comparator)
  Interventions: Procedure: inverted flap
- peeling internal limiting membrane (ILM) (Active Comparator)
  Interventions: Procedure: peeling internal limiting membrane (ILM)

INTERVENTIONS:
Procedure: inverted flap — full thickness macular hole surgery
  Arms: inverted flap
Procedure: peeling internal limiting membrane (ILM) — full thickness macular hole surgery
  Arms: peeling internal limiting membrane (ILM)

SUMMARY:
Primary outcome: difference of microperimetry retinal sensitivity after primary vitrectomy for idiopathic full thickness macular holes with inverted flap technique versus internal limiting membrane (ILM) peeling technique Secondary outcomes: difference of visual change after primary vitrectomy for idiopathic full thickness macular holes with inverted flap technique versus internal limiting membrane (ILM) peeling technique; difference in closure rate after primary vitrectomy for idiopathic full thickness macular holes with inverted flap technique versus internal limiting membrane (ILM) peeling technique

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* idiopathic full thickness macular hole ≤ 350 micron of diameter
* phakic or pseudophakic
* absence of systemic adverse conditions

Exclusion Criteria:

* concomitant retinal and other ocular disease
* previous ocular surgery except cataract surgery
* axial length >26mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Microperimetry retinal sensitivity | 3 months
  Difference of microperimetry retinal sensitivity after primary vitrectomy for idiopathic full thickness macular holes with inverted flap technique versus internal limiting membrane (ILM) peeling technique

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) | 3 months
  Difference of best corrected visual acuity (BCVA) after primary vitrectomy for idiopathic full thickness macular holes with inverted flap technique versus internal limiting membrane (ILM) peeling technique
Closure rate | 3 months
  Closure rate after primary vitrectomy for idiopathic full thickness macular holes with inverted flap technique versus internal limiting membrane (ILM) peeling technique

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U. Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ventre L, Fallico M, Longo A, Parisi G, Russo A, Bonfiglio V, Marolo P, Caselgrandi P, Avitabile T, Borrelli E, Reibaldi M. CONVENTIONAL INTERNAL LIMITING MEMBRANE PEELING VERSUS INVERTED FLAP FOR SMALL-TO-MEDIUM IDIOPATHIC MACULAR HOLE: A Randomized Trial. Retina. 2022 Dec 1;42(12):2251-2257. doi: 10.1097/IAE.0000000000003622. Epub 2022 Sep 6. PMID 36084331